CLINICAL TRIAL: NCT00452114
Title: A Randomized, Controlled Study Evaluating the Effectiveness of the Inexsufflator Cough Assist Device in Patients With Symptomatic Bronchiectasis
Brief Title: In-exsufflator Cough Assist Device in Patients With Symptomatic Bronchiectasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis indicates statistical futility for primary outcomes
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Stephen Krinzman, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-11138
Record Dates: First submitted 2007-03-22; First posted 2007-03-26 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Assignment to In-Exsufflator Cough Assist Device (Active Comparator): In-Exsufflator Cough Assist Device augments the expiratory flow and force of the patient's cough with the addition of a cycle of positive and negative inspiratory pressure when used daily
  Interventions: Device: In-Exsufflator Cough Assist Device
- Assignment to flutter valve device (Active Comparator): flutter valve device delivers expiratory low-pressure vibratory pulse to the patient's airway when used daily
  Interventions: Device: Active Comparator: Flutter Valve Device

INTERVENTIONS:
Device: In-Exsufflator Cough Assist Device
  Arms: Assignment to In-Exsufflator Cough Assist Device
Device: Active Comparator: Flutter Valve Device — Active Comparator
  Arms: Assignment to flutter valve device

SUMMARY:
This study is a randomized, controlled trial examining the effectiveness of the mechanical cough-assist device (in-exsufflator) in promoting the clearance of retained airway secretions in patients with symptomatic bronchiectasis. We hypothesize that this enhanced clearance of airway secretions will lead to a decline in the number of acute exacerbations of bronchiectasis experienced by these patients during the study period, improve health-related quality of life, decrease overall health-care costs and improve pulmonary function.

DETAILED DESCRIPTION:
Bronchiectasis is characterized by airway dilatation with the potential to cause devastating illness, including repeated respiratory infections requiring antibiotics, disabling productive, mucopurulent cough, shortness of breath and occasional hemoptysis. The damaged and dilated airways lead to persisting bacterial infection of the bronchi and bronchioles, causing inflammation and retained secretions, which in turn may further damage the airways. Patients typically suffer from frequent, severe and refractory episodes of bacterial bronchitis, often requiring hospitalization and prolonged courses of antibiotics. The pathophysiology of bronchiectasis involves the retention of viscid, tenacious inflammatory secretions and microbes leading to a "vicious cycle" of airway obstruction, destruction and recurrent infection with further compromise of the mucociliary clearance host defense apparatus. It has been widely proposed and recommended that methods of enhancing clearance of airway secretions should be an integral component of the care of patients with bronchiectasis. Despite these recommendations and a sound pathophysiologic plausibility given the central role retention of secretions plays in the disease, the effectiveness of interventions targeted toward enhancing bronchopulmonary hygiene has not been systematically studied. It is also not known whether the ability to generate an adequate cough would predict which patient will benefit from these interventions.

The mechanical in-exsufflator device assists patients in clearing retained secretions by augmenting the expiratory flow and force of the patient's cough with the addition of a cycle of positive and negative inspiratory pressure. An effective cough mechanism is actually an important and beneficial host defense which aids in mucus clearance along with the mucociliary apparatus. We hypothesize that daily, regular use of the in-exsufflator device will lead to a reduction in acute bronchiectasis exacerbations- a clinically meaningful endpoint- with other possible beneficial outcomes including improved pulmonary function, improved health-related quality of life and decreased health care costs.

Despite the lack of rigorous, well-designed studies supporting the role and most effective mode of bronchial hygiene physiotherapy in patients with bronchiectasis, many Pulmonologists recommend the flutter valve device as the generally accepted "standard of care" at this time due to its relative non-invasiveness, ease of use and high level of patient acceptability. The flutter valve is a simple, hand-held, pipe-like device which helps loosen secretions by providing an expiratory low-pressure vibratory pulse to the patient's airway when used. This study will provide a comparison of the clinical efficacy of these mechanical chest physiotherapy devices in the setting of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Chest CT scan confirmation of bronchiectasis
* At least two exacerbations in the preceding 12 months requiring antibiotics

Exclusion Criteria:

* Cystic fibrosis
* Bullous emphysema
* History of spontaneous pneumothorax
* History of massive hemoptysis: greater than 200 cc in a 24 hour period
* Lung resection surgery in the past 6 months
* Use of the mechanical cough in-exsufflator in the prior 3 months
* Inability to speak and read English
* Inability to demonstrate proper use of the cough-assist or flutter device
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Krinzman, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - UMass Memorial Medical Center, Universty Campus, Worcester, Massachusetts
  - St. Vincent Medical Center, Worcester, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- In-Exsufflator Cough Assist Device: In-Exsufflator Cough Assist Device augments the expiratory flow and force of the patient's cough with the addition of a cycle of positive and negative inspiratory pressure when used daily
- Flutter Valve Device: flutter valve device delivers expiratory low-pressure vibratory pulse to the patient's airway when used daily
Period: Overall Study
Arm/Group | In-Exsufflator Cough Assist Device | Flutter Valve Device
Started | 15 | 13
Completed | 12 | 10
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Exsufflator Cough Assist Device | Flutter Valve Device | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Suppurative Exacerbations Per Patient Per Year
Description: The impact of the intervention is measured by the total number of suppurative exacerbations per patient within a 12 month period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of events per patient
Arm/Group | Participants in the Intervention Group (Cough In-exsufflator) | Particpants in the Control Group (Flutter Device)
Number analyzed (Participants) | 12 | 10
Number of events per patient | 2.5 (1.7) | 2.3 (2.1)

2. Primary Outcome: Number of Hospitalizations and Urgent/Unscheduled Outpatient Visits
Description: The impact of the intervention is measured by the number of hospitalizations and urgent/unscheduled outpatient visits the participants experienced within a 12 month period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Hospitalizations/Visits
Arm/Group | Participants in the Intervention Group (Cough In-exsufflator) | Particpants in the Control Group (Flutter Device)
Number analyzed (Participants) | 12 | 10
Number of Hospitalizations/Visits | .78 (.8) | .87 (1.2)

3. Secondary Outcome: Quality of Life (St. George's Respiratory Questionnaire)
Description: Quality of life is measured using St. George's Respiratory Questionnaire, a 50 item disease-specific instrument designed to measure impact on overall health, daily life and perceived well-being in patients with obstructive airways disease. The instrument consists of 2 parts, and 3 components. Part 1 measures symptom frequency and severity with a 1,3 or 12 month recall. Part 1 is evaluated using several scales. Part 2 measures impact of breathlessness on activities including social functioning and psychological disturbances. Part 2 is evaluated by dichotomous (true false) evaluation except the final question which is a 4 point likert scale. Scores range from 0 to 100 with higher score indicating more limitation and lower quality of life.
Time Frame: 12 months
Population: Outcomes not analyzed
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Participants in the Intervention Group (Cough In-exsufflator) | Particpants in the Control Group (Flutter Device)
Number analyzed (Participants) | 12 | 10
scores on a scale | 30 (14) | 24 (9)

4. Secondary Outcome: Quality of Life (Cough-Specific Quality of Life Questionnaire)
Description: Quality of life is measured using the Cough Specific Quality of Life Questionnaire (CQLQ) to measure the effect of interventions on cough-specific quality of life. The Cough-Specific Quality of Life Questionnaire consist of 28 questions about cough and its effects using Likert-like 4-point scales, with lower scores indicating less effect of cough on health related quality of life.
  CQLQ scale ranges from 28 to 112 with higher scores indicating worse outcome or status.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants in the Intervention Group (Cough In-exsufflator) | Particpants in the Control Group (Flutter Device)
Number analyzed (Participants) | 12 | 10
Scores on a scale | 48 (15) | 43 (10)

ADVERSE EVENTS:
Arm/Group | In-Exsufflator Cough Assist Device | Flutter Valve Device
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Study terminated due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes